CLINICAL TRIAL: NCT03401151
Title: Changes in Skeletal Muscle Over Time in Severe Heart Failure
Brief Title: CHANges iN skEletal muscLe in Heart Failure
Acronym: Channel-HF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Thomas Gustafsson Assoc Prof, Professor, Karolinska Institutet
Other Study IDs: Channel-HF KI
Record Dates: First submitted 2017-11-20; First posted 2018-01-17 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Heart Failure
Keywords: Heart failure; Skeletal muscle; Exercise capacity; Lung function; Gene expression
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples, muscle biopsies
  Initial examination and sampling:
  A) Blood sampling B) Ecocardiographic examination, C) Maximal working test including oxygen uptake D) Measurement of arm and leg strength using so-called Biodex E) Pulse, blood pressure and cardiac output volume measurement F) Measurement of muscle mass using CT G) Muscle biopsy in local anesthesia taken from one leg's vastus lateralis H) Daily physical activity measured with an accelerometer (pedometer) I) Measurement of lung function using standard spirometry J) Cardiac examination with MR in non-pacemaker subjects
  24 months after the first sampling, the persons will be asked to re-examine the same examination procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The mechanisms behind heart failure are largely unknown. Despite an increasing arsenal of pharmacological therapies, cardiovascular disease is still the most common cause of death in the western world, which demonstrates a pronounced need for more patient-related mechanistic research. Cachexia and limited exercise capacity are the symptoms that best match prediction of heart failure, both of which are symptoms involving a dysfunctional skeletal muscle. An increased understanding of the mechanisms and signaling pathways connects the failure heart with skeletal muscle dysfunction is likely to lead both to discoveries of prognostic factors and possible therapeutic options.

The study is a prospective, non-blinded, study. The study will consist of the assignment of patients with heart failure, New York Heart Association (NYHA) III-IV, 60-80 years old. One hundred (100) patients will be enrolled in this study.

DETAILED DESCRIPTION:
The primary objective is to investigate how changes in the skeletal muscle coincide with changes in physical performance, cardiac function, and prognosis in patients with heart failure, and changes over time. Therefore, the investigators will investigate patients with severe heart failure at 'baseline' and on a second follow-up occasion after 12-16 months.

The secondary and tertiary objective is to investigate how changes in the metabolic signature of blood and satellite cells coincide with changes in physical performance, cardiac function, and prognosis in patients with heart failure, and changes over time. Patient recruitment is expected to occur over 36 months.

The study will be conducted in Sweden at Karolinska University Hospital, Huddinge.

ELIGIBILITY:
Inclusion criteria:

* Signed informed consent
* 60-80 years old upon inclusion
* Chronic heart failure ≥ 45 days.
* Left ventricular ejection fraction ≤ 35%.
* NYHA III-IV
* Receiving medical management with optimal doses of betablockers, acetylcholinesterase (ACE)-inhibitors or angiotensin II receptor blockers (ARB), and mineral receptor antagonists (MRA) for at least 30 days if tolerated.

Exclusion criteria:

* Interagency Registry for Mechanically Assisted Circulatory Support (INTERMACS) profile 1 "crash and burn"
* On-going mechanical circulatory support.
* Severe chronic obstructive pulmonary disease (COPD) or severe restrictive lung disease.
* Psychiatric disease, cognitive dysfunction, alcohol or drug abuse, or psychosocial issues that are likely to impair study compliance
* Condition, other than heart failure, requiring end-of-life care within <6 months in time or where the risk of death within <2 years is considered to be imminent.
* Participation in studies that resulted in departure from normal treatment routine or invasive investigations within <6 months back in time.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe heart failure
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Metabolic signature of muscle, messenger RNA (mRNA) gene expression | Change from baseline metabolic signature at 24 months
  Metabolomics profile using nuclear magnetic resonance (NMR)
Metabolic signature of muscle, messenger RNA (mRNA) gene | Change from baseline metabolic signature at 24 months
  Metabolomics profile using liquid chromatography-high-resolution mass spectrometry (LC-HRMS)

SECONDARY OUTCOMES:
Metabolic signature of blood, mRNA gene expression | Change from baseline metabolic signature at 24 months
  Metabolomics profile using NMR
Metabolic signature of blood, mRNA gene expression | Change from baseline metabolic signature at 24 months
  Metabolomics profile using LC-HRMS
Metabolic signature of satellite cells, mRNA gene expression | Change from baseline metabolic signature at 24 months
  Metabolomics profile using NMR
Metabolic signature of satellite cells, mRNA gene expression | Change from baseline metabolic signature at 24 months
  Metabolomics profile using LC-HRMS
Expression levels of targeted genes using transcriptomics | Change from baseline metabolic signature at 24 months
  Choice of genes based on results obtained by metabolomics approaches

CONTACTS AND LOCATIONS:
Overall Officials: Matti Sällberg, professor, Study Chair — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided